CLINICAL TRIAL: NCT01339546
Title: National Trends In Ambulatory Care Visits For Otitis Media In Children Under The Age Of Five In The United States
Brief Title: National Trends in Otitis Media in Children Under 5 Years of Age
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 6096A1-4018; B1851041 (Other: Alias Study Number)
Record Dates: First submitted 2010-12-22; First posted 2011-04-20 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2017-11

CONDITIONS: Otitis Media; Myringotomy Tube Insertion; Skin Rash; Trauma
Keywords: ecologic; cross sectional; trend analysis
MeSH Terms: conditions — Otitis Media; Exanthema; Wounds and Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: All ambulatory visits for otitis media, myringotomy tube insertion, skin rash or trauma among children age 5 or under during the periods of study
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The rationale for this study is to assess the change in ambulatory care visit rates for acute otitis media between the period before (2001-2009) and after the introduction of the 13-valent pneumococcal conjugate vaccine (13vPnC) (2011-2013) among children less than 5 years old in the United States.

DETAILED DESCRIPTION:
NAMCS-The survey utilizes a three stage sampling design based on (1) probability of selecting a primary sampling unit (PSU) (2) probability of selecting a physician within the PSU and (3) probability of selecting a patient within the physician practice. This last probability is defined to be the exact number of office visits during physician's specified reporting week divided by the number of patient record forms completed. NHAMCS- For producing unbiased national estimate, this survey utilizes four stages (a) Probability of selecting a PSU (b) probability of selecting a hospital with in PSU (c) probability of selecting an emergency department (ED) or outpatient department (OPD) within the hospital (d) probability of selecting a visit within ED or OPD. The overall probability of selection is the product of the probabilities at each stage. The inverse of the overall selection probability is the basic inflation weight.

ELIGIBILITY:
Inclusion Criteria:

Five years of age or under at the time of visit, ambulatory visit for otitis media, myringotomy tube insertion, skin rash or trauma during study period

Exclusion Criteria:

Age over 5 years, no ambulatory visits for the events listed in inclusion criteria

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: National Ambulalatory Medical Care Survey (NAMCS)-national sample of visits to non federally employed office based physicians who are primarily engaged in direct patient care, and National Hospital Ambulatory Medical Care Survey (NHAMCS)- national sample of visits to emergency and outpatient departments and to ambulatory surgery facilities in noninstitutional general and short stay hospitals, exclusive of Federal, military, and Veterans Administration hospitals, located in the 50 States and the District of Columbia
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory care visit rates for acute otitis media between the period before (2001-2009) and after the introduction of the 13vPnC vaccine (2011-2013) among children less than 5 years old | 1) 2001-2009 inclusive (9 years) and 2) 2011-2013 inclusive (3 years)

SECONDARY OUTCOMES:
Change in ambulatory care visit rates for acute otitis media between: 1) 1997-99 to 2001-09; and 2) between 1997-99 to 2011-13 among children less than 5 years old. (Timeframes are retrospective) | 1) 1997-99 inclusive (3 yrs); 2) 2001-09 inclusive (9 yrs) and 3) 2011-13 inclusive (3 yrs)
Change in ambulatory care visit rates for myringotomy tube insertion between: 1) 1997-99 to 2001-09; and 2) between 1997-99 to 2011-13 among children less than 5 years old. (Timeframes are retrospective | 1) 1997-99 inclusive (3 yrs); 2) 2001-09 inclusive (9 yrs) and 3) 2011-13 inclusive (3 yrs)
Change in ambulatory care visit rates for rash between 2001-09 to 2011 -13 among children less than 5 years old. (Timeframes are retrospective) | 1) 2001-09 inclusive (9 yrs) and 2) 2011-13 inclusive (3 yrs)
Change in ambulatory care visit rates for trauma between 2001-09 to 2011-13 among children less than 5 years old. (Timeframes are retrospective) | 1) 2001-09 inclusive (9 yrs) and 2) 2011-13 inclusive (3 yrs)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-4018&StudyName=National%20Trends%20in%20Otitis%20Media%20in%20Children%20Under%205%20Years%20of%20Age%20